CLINICAL TRIAL: NCT01373619
Title: Heart Failure With Normal Ejection Fraction (HFNEF) in Hemodialysed Patients: Beneficial Effect of Ivabradine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Gennaro Cice, MD Second University of Naples, Second University of Naples
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HFNEF-IVA-DIAL
Record Dates: First submitted 2011-05-25; First posted 2011-06-15 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2010-01

CONDITIONS: Heart Failure
Keywords: Heart failure with normal ejection fraction; hemodialysis patients; ivabradine; Echocardiography; NYHA class; 6-minutes walking test
MeSH Terms: conditions — Heart Failure | interventions — Ivabradine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IVABRADINE, HEART FAILURE WITH NORMAL EF (Experimental): Patient on hemodialysis with Heart failure with normal ejection fraction treated with ivabradine titrated to 7.5 mg BID to assess changes in echocardiography diastolic function and NYHA class and 6-minutes walking test
  Interventions: Drug: Ivabradine

INTERVENTIONS:
Drug: Ivabradine — ivabradine titrated to 7.5 mg BID
  Other Names: Procoralan; Corlentor

SUMMARY:
Heart failure with normal ejection fraction is often under diagnosed and certainly under treated in hemodialyzed patients. Because of the benefit of reducing heart rate, ivabradine, a pure heart-rate lowering agent without effects on blood pressure, is of potential therapeutic utility.

ELIGIBILITY:
Inclusion Criteria:

* hemodialyzed patients
* signs and symptoms of heart failure with normal ejection fraction
* sinus rhythm

Exclusion Criteria:

* atrial fibrillation/atrial flutter
* valvular heart disease
* unstable angina
* hospitalization for heart failure prior 3 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Echocardiofic changes of diastolic left ventricular function | baseline, 1, 3, 6, 9, 12 months
  Measures of diastolic left ventricular function (E and A velocity and deceleration time of mitral inflow and Doppler-Tissue-Imaging E velocity and their ratio) were assessed at baseline and at each scheduled time.

SECONDARY OUTCOMES:
changes in NYHA class | baseline, 1,3,6,9,12 months
  Measures of New York Heart Association functional class stratified I to IV at baseline and at each scheduled time.
changes in 6-minutes walking test | baseline, 1,3,6,9,12 months
  American Thoracic Society At baseline and at each scheduled time a 6-minutes walking test were performed according ATS Statement. The following measures were analysed at starting and ending test: heart rate; blood pressure, dyspnea according the Borg scale, fatigue according the Borg scale, Spo2%;distance walked, symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Gennaro Cice, MD, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Chair of Cardiology Second Univesity of Naples, Naples, Italy